CLINICAL TRIAL: NCT07034807
Title: Evidence-based Evaluation of Yiqi Jiangzhuo Huoxue Tongluo Method in Delaying the Occurrence of End-stage Renal Disease in Diabetic Kidney Disease--Study 2
Brief Title: YiqiJiangzhuoHuoxueTongluo Method to Delay the Occurrence of End-stage Renal Disease in Diabetic Kidney Disease--Study2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Hongfang (Other)
Collaborators: Guang'anmen Hospital，China Academy of Chinese Medical Sciencescancel (Unknown); First Affiliated Hospital, Sun Yat-Sen University (Other); Tianjin Medical University Chu Hsien-I Memorial Hospital (Unknown); The Affiliated Hospital to ChangChun University of Chinese Medicinecancel (Unknown); EFONG PHARMRCEUTICRL (Unknown)
Responsible Party: Sponsor-Investigator, Liu Hongfang, Chief Physician, Dongzhimen Hospital, Beijing
Organization: Dongzhimen Hospital, Beijing (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023ZD0509303-2
Record Dates: First submitted 2025-04-08; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Kidney Disease (DKD)
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: the practical randomized controlled trial designed by Zelen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shenzhuo Decoction (Experimental): The experimental group was given the traditional Chinese medicine prescription ' Shenzhuo Decoction ' ( composed of Astragalus membranaceus, Salvia miltiorrhiza, Leech, Raw Rhubarb, Epimedium, Motherwort ) + basic treatment ( including nutrition, lifestyle, hypoglycemic, hypotensive, lipid-lowering, control of other risk factors, etc. )
  Interventions: Drug: the traditional Chinese medicine prescription ' Shenzhuo Decoction '; Combination Product: basic treatment
- basic treatment (Active Comparator): the control group was given basic treatment, a total of 1 year of drug intervention（including nutrition, lifestyle, hypoglycemic, hypotensive, lipid-lowering, control of other risk factors, etc.）
  Interventions: Combination Product: basic treatment

INTERVENTIONS:
Drug: the traditional Chinese medicine prescription ' Shenzhuo Decoction ' — The traditional Chinese medicine prescription ' Shenzhuo Decoction ' is composed of Astragalus membranaceus, Salvia miltiorrhiza, Leech, Raw Rhubarb, Epimedium, Motherwort. It is a traditional Chinese medicine prescription for the treatment of diabetic kidney disease, which was founded by Tong Xiaolin, an academician of the Chinese Academy of Sciences.
  Other Names: Chinese medicine
  Arms: Shenzhuo Decoction
Combination Product: basic treatment — Basic treatment includes six aspects : nutrition, lifestyle, hypoglycemic, hypotensive, lipid-lowering, and control of other risk factors, which are implemented in accordance with clinical standard treatment specifications.
  Other Names: control group

SUMMARY:
Using the practical randomized controlled trial designed by Zelen, the subjects were randomly divided into the experimental group and the control group. The experimental group was given the traditional Chinese medicine prescription ' Shenzhuo Decoction ' ( composed of Astragalus membranaceus, Salvia miltiorrhiza, Leech, Raw Rhubarb, Epimedium, Motherwort ) + basic treatment ( including nutrition, lifestyle, hypoglycemic, hypotensive, lipid-lowering, control of other risk factors, etc. ), the control group was given basic treatment, a total of 1 year of drug intervention, followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* 1 In line with the diagnostic criteria of Western medicine type 2 DKD ;
* 2 18-80 years old, regardless of gender ;
* 3 30ml / min / 1.73m2 ≤ eGFR < 60ml / min / 1.73m2 ( eGFR was calculated according to CKD-EPI formula ) ;
* 4 In line with the diagnostic criteria of qi deficiency and collateral stasis syndrome in traditional Chinese medicine ;
* 5 hbA1c between 7-10 % ;
* 6 uACR ≥ 300mg / g
* 7 blood pressure ≤ 150 / 90mmHg ;
* 8 signed the informed consent ;

Exclusion Criteria:

* 1 Patients who are currently receiving other traditional Chinese medicines and Chinese patent medicines with DKD therapeutic effects ;
* 2 combined with other clear renal diseases, such as polycystic kidney disease, glomerulonephritis, renal tumors ;
* 3 Patients with acute or chronic infection who needed treatment were judged by the researchers not suitable for inclusion in the study ;
* 4 Patients who participated in any other research drug study and / or received or had received another research drug or intervention treatment ( within one month before signing the informed consent form ) ;
* 5 patients who were allergic or contraindicated to the planned use of drugs ;
* 6 There are serious acute or chronic diseases that the major researchers believe may pose an excessive risk to the subjects, including : patients with cardiovascular, cerebrovascular, lung, blood, digestive tract, liver, kidney, neuropsychiatric or infectious diseases ;
* 7 Patients with a history of immunodeficiency, including patients with other acquired, congenital immunodeficiency diseases, or patients with a history of organ transplantation or planned organ transplantation ;
* 8 Women with positive pregnancy screening test or lactating or planning to get pregnant in the next 24 months. Female or male patients who were reluctant to use contraception throughout the study period ;
* 9 patients with a history of malignant tumors within 5 years ;
* 10 patients with type 1 diabetes ;
* 11 patients with maintenance dialysis > 2 weeks and / or expected maintenance dialysis > 8 weeks before treatment and patients who were judged by any researcher not suitable for inclusion in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate ( eGFR ) decline slope | At the time of enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.

SECONDARY OUTCOMES:
The incidence of renal composite outcome | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Defined as the occurrence of end-stage renal disease [ dialysis, transplantation or glomerular filtration rate ( eGFR ) < 15ml / ( min · 1.73m2 ) ], eGFR decreased by more than 50 %, death caused by renal causes
Urinary albumin creatinine ratio (UACR ) | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
Changes in 24-hour urinary protein levels | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
Estimate the change value of glomerular filtration rate ( eGFR ) level, slope | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
Changes of Traditional Chinese Medicine syndrome integrals | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  The symptoms of the patients were scored with the Traditional Chinese Medicine syndrome scale to better judge the changes of the symptoms of the patients.The highest score was 114 points, and the lowest score was 0 points. The higher the score, the worse the patient 's health.

OTHER OUTCOMES:
Body temperature | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
blood pressure | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Both systolic and diastolic blood pressures should be measured
respiration | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
heart rate | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
Number of participants with abnormal white blood cell count ( WBC ) | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal white blood cell count ( WBC )
Number of participants with abnormal red blood cell count ( RBC ) | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal red blood cell count ( RBC )
Number of participants with abnormal electrocardiogram | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal electrocardiogram
Number of participants with abnormal hemoglobin ( HGB ) | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal hemoglobin ( HGB )
Number of participants with abnormal lymphocyte percentage ( LY % ) | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal lymphocyte percentage ( LY % )
blood lipid | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
glycosylated hemoglobin | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
fasting blood glucose | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
incidence of adverse events | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
Number of participants with abnormal Percentage of neutrophils( NE % ) | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Percentage of neutrophils( NE % )
Number of participants with abnormal Platelet count ( PLT ) | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Platelet count ( PLT )
Number of participants with abnormal Urine PH value | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Urine PH value
Number of participants with abnormal Urinary protein | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Urinary protein
Number of participants with abnormal Urine occult blood | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Urine occult blood
Number of participants with abnormal Urinary glucose | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Urinary glucose
Number of participants with abnormal Urine ketone | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Urine ketone
Number of participants with abnormal Urine white blood cells (high magnification field of view) | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Urine white blood cells (high magnification field of view)
Number of participants with abnormal Urine red blood cells (high magnification field of view) | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Urine red blood cells (high magnification field of view)
Number of participants with abnormal Serum alanine aminotransferase | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Serum alanine aminotransferase
Number of participants with abnormal Serum aspartate aminotransferase | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Serum aspartate aminotransferase
Number of participants with abnormal Serum alkaline phosphatase | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Serum alkaline phosphatase
Number of participants with abnormal Serum gamma-glutamyl transferase | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Serum gamma-glutamyl transferase
Number of participants with abnormal Serum albumin (ALB) | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Serum albumin (ALB)
Number of participants with abnormal Serum total bilirubin（TBIL） | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Serum total bilirubin（TBIL）
Number of participants with abnormal Serum direct bilirubin（DBIL） | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Serum direct bilirubin（DBIL）
Number of participants with abnormal Serum indirect bilirubin （IBIL） | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Number of participants with abnormal Serum indirect bilirubin （IBIL）
Serum urea | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Serum urea
Serum urate | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Serum urate
Serum cystatin C | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Serum cystatin C
Serum creatinine | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Serum creatinine
Plasma triglyceride | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Plasma triglyceride
Plasma high-density lipoprotein | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Plasma high-density lipoprotein
Plasma low-density lipoprotein | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Plasma low-density lipoprotein
Plasma total cholesterol | Introduction period ( 1 month before enrollment ), enrollment, 6 months ± 1 week, 12 months ± 1 week, 18 months ± 1 week, 24 months ± 1 week after enrollment.
  Plasma total cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: HongFang Liu, Study Director — Dongzhimen Hospital
Locations (5):
- China (5):
  - Dongzhimen Hospital, Beijing, Beijing Municipality
  - Guang'anmen Hospital，China Academy of Chinese Medical Sciencescancel, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Affiliated Hospital to ChangChun University of Chinese Medicinecancel, Changchun, Jilin
  - Tianjin Medical University Chu Hsien-I Memorial Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No